CLINICAL TRIAL: NCT01889355
Title: User Study for the Evaluation of an Enhanced Meter Feature Using an AgaMatrix BGMS
Brief Title: User Study for Enhanced Meter Feature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AgaMatrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AGAFPGM01
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2014-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; glucose; glucometer
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enhanced meter feature usability (Other): Home diabetes monitoring by patient using provided blood glucose monitoring system.
  Interventions: Device: AgaMatrix Blood Glucose Monitor

INTERVENTIONS:
Device: AgaMatrix Blood Glucose Monitor

SUMMARY:
This enhanced meter feature raises awareness among patients by providing additional information regarding their glycemic control in between Healthcare Professional visits. This information may facilitate increased dialogue between patient and Healthcare Professional and can remind patients of the importance of glycemic control.

This study will evaluate a user's ability to use the enhanced meter feature.

ELIGIBILITY:
Inclusion criteria:

IC 1. Age of subject is 18 years or older

IC 2. Type I or type II diabetes inclusive of the following populations:

1. Mixed insulin therapies
2. Basal insulin therapies
3. Bolus insulin therapies
4. CSII therapies
5. MDI therapies
6. Non-insulin diabetic treatments (oral and injectable)
7. Life style (exercise and diet) diabetes management IC 3. Able to speak and read English proficiently

Exclusion criteria EC 1. Pregnant EC 2. Hct <20 or >60 EC 3. Work for BGM competitor company (including, but not limited to Lifescan, Roche, Abbott) EC 4. Homeless EC 5. Incarcerated EC 6. Institutionalized EC 7. Employees or students of the Research Site, including the Principal Investigator, directly involved in the conduct of the protocol.

EC 8. Has any condition that the Principal Investigator believes may interfere in the subject's participation in the study.

EC 9. Previous experience using the MyStar Extra BGMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta Diabetes Associates, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Procedure: 5.5 Evaluation Procedure The evaluation shall be performed in the following sequence and be supervised by one or more healthcare providers trained in the use of the device under evaluation (ISO 15197:2013 8.1).
  1. Briefly describe to the subject that the goal of this study is to obtain a blood glucose reading, describe the study procedures, and obtain written informed consent ensuring all questions are answered.
  2. For each consenting study subject, assign a sequential User ID number and obtain inclusion criteria, exclusion criteria, and user demographics.
  3. Perform a urine pregnancy test for women of childbearing potential if pregnancy status unknown.
  4. Locate subjects to a private area where they are not able to see others performing the test.
  5. The trained technician will put on a new pair of gloves.
  6. Provide the subject with an AgaMatrix meter, test strips, the system kit lancing device and lancets. Prior to performing self-testing, each study subject shall
Period: Overall Study
Arm/Group | Study Procedure
Started | 115
Completed | 113
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Demographics: Age group ranged from ages 18-86, Male and female with both Type 1 and Type 2 diabetics. Race was both white, black/African American and Hispanic who are able to read and understand English per the subject consent form.
Arm/Group | Demographics
Number analyzed (Participants) | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 107
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Enhanced Meter Feature Usability
Description: The primary objective of this study is to evaluate that the intended users are able to obtain accurate blood glucose measurements when operating the blood glucose monitoring system, given only the training materials routinely provided with the system (ISO 15197:2013 8.1).
Time Frame: 4 weeks
Population: All diabetic subjects who volunteer for the study and qualify in accordance with the study inclusion and exclusion criteria, the user requirements established by the manufacturer for the blood-glucose system, and applicable regulatory requirements, shall be eligible to participate in the study
Measure: Count of Participants; unit: Participants
Groups:
- Subject Population, Inclusion and Exclusion: This clinical study will consist of at least 50 evaluable subjects who meet all inclusion/exclusion criteria.
  Subjects shall be selected using the consecutive sampling method. All diabetic subjects who volunteer for the study and qualify in accordance with the study inclusion and exclusion criteria, the user requirements established by the manufacturer for the blood-glucose system (e.g. packed cell volume within the system's specified limits), and applicable regulatory requirements (e.g. written informed consent), shall be eligible to participate in the study (ISO 15197:2013 8.3).
  3.2 Inclusion Criteria
  Potential participants may be enrolled in the study if they satisfy the following inclusion criteria:
  IC 1. Age of subject is 18 years or older IC 2. Has been diagnosed with Type1 or Type 2 diabetes IC 3. Able to speak and read English proficiently IC 4. Must be physically able to self-test
  3.3 Exclusion Criteria Potential subjects who display any o
Arm/Group | Subject Population, Inclusion and Exclusion
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Groups:
- Adverse and Serious Events: No adverse or serious events occurred during this study
Arm/Group | Adverse and Serious Events
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No